CLINICAL TRIAL: NCT02363855
Title: An Open Label Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BAY 1841788 in Japanese Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: Phase 1 Dose Escalation Study of BAY 1841788 in Japanese Metastatic Castration-resistant Prostate Cancer (mCRPC) Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17719
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Prostatic Neoplasms
Keywords: Neoplasm Metastasis; Metastatic castration-resistant prostate cancer; Castration-resistant prostate cancer (CRPC)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BAY 1841788(ODM-201) (Experimental): Cohort 1: Safety, tolerability and PK of 300 mg dose given twice daily. Escalation to cohort 2 in case no safety relevant adverse event has been observed within 28 days after start of multiple dose (MD) Cohort 2: Safety, tolerability and PK of 600 mg dose given twice daily
  Interventions: Drug: BAY 1841788(ODM-201)

INTERVENTIONS:
Drug: BAY 1841788(ODM-201) — Cohort 1: Single dose 300 mg BAY 1841788, followed by twice daily administration of the same dose for 12 weeks Cohort 2: Single dose 2x300 mg BAY 1841788, followed by twice daily administration of the same dose for 12 weeks.

SUMMARY:
The primary objectives of this study are to investigate the safety and tolerability of BAY 1841788 in Japanese subjects with metastatic castration-resistant prostate cancer (mCRPC) and the PK of BAY 1841788 and its major metabolite BAY 1896953.

DETAILED DESCRIPTION:
The drug product is licensed from Orion pharma, Finland which is also the manufacturer of the product.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males aged ≥ 20 years
* Histologically or cytologically confirmed adenocarcinoma of prostate without neuroendocrine differentiation or small cell features
* Patients with metastatic castration-resistant prostate cancer (mCRPC). CRPC is defined as follows

  * Ongoing androgen deprivation therapy with a luteinizing hormone-releasing hormone (LHRH) analogue or antagonist, or bilateral orchiectomy, and castrate level of serum testosterone (< 1.7 nmol/l [50 ng/dL]) at screening AND
  * Progressive disease and/or prostate-specific antigen (PSA) increase of three consecutive rises, at least 1 week apart AND
  * PSA > 2ng/mL at screening
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1
* Life expectancy of at least 3 months
* Blood counts at screening: haemoglobin ≥ 9.0 g/dL, absolute neutrophil count ≥ 1,500/μL (1.5x109/l), platelet count ≥ 100,000/μL (100x109/l) (patient must not have received any growth factor or blood transfusion within 7 days of the hematology laboratory obtained at screening)
* Screening values of serum alanine aminotransferase (ALT) and/or aspartate transaminase (AST) ≤ 2.5 x upper limit of normal (ULN), total bilirubin ≤ 1.5 x ULN, creatinine ≤ 1.5 x ULN, albumin > 3.0 g/dl
* Prior treatment with antiandrogen. Discontinuation of bicalutamide or nilutamide (not approved in Japan) at least 6 weeks and other antiandrogens at least 4 weeks prior to the start of the study drug administration.

Exclusion Criteria:

* Known metastases in the brain
* Symptomatic local-regional disease that requires medical intervention including moderate/severe urinary obstruction or hydronephrosis due to prostate cancer
* Acute toxicities (except for alopecia and CTCAE grade 2 neuropathy) of prior treatments and procedures not resolved to CTCAE ≤ grade 1 or baseline before the first drug administration
* Febrile neutropenia of Common Terminology Criteria for Adverse Events (CTCAE) ≥ 3
* History of other malignancy within the previous 5 years except a basal cell carcinoma of skin and any other cancer for which treatment has been completed ≥ 5 years ago and from which the patient has been disease-free5 years ago and from which the patient has been disease-free
* Prior treatment within 4 weeks before the first drug administration with immunotherapy, antiandrogen, CYP17 inhibitor (CYP17i), oral ketoconazole, estrogens, 5-α reductase inhibitors or investigational treatment
* Use of bicalutamide or nilutamide (not approved in Japan) within 6 weeks before the first drug administration
* Radiation therapy (external beam radiation therapy [EBRT], brachytherapy, or radiopharmaceuticals) or chemotherapy (except for nitrosoureas and mitomycin C) within 4 weeks before the first drug administration. Use of nitrosoureas or mitomycin C within 6 weeks before the first drug administration.
* Prior use of any herbal products known to decrease PSA levels (e.g. PC SPES or saw palmetto) within 4 weeks before the first drug administration

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Event as measure of safety and tolerability | Up to 12 weeks
The intensity of an adverse event graded using the NCI CTCAE version 4.03 | Up to 12 weeks
  National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE)
Plasma concentration of BAY 1841788 characterized by Cmax | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  Cmax: maximum drug concentration in plasma after single dose administration
Plasma concentration of BAY 1841788 characterized by tmax | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  tmax: time to reach maximum drug concentration in plasma after single (first) dose
Plasma concentration of BAY 1841788 characterized by AUC(0-12) | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  AUC(0-12):AUC from time 0 to 12 hours after administration
Plasma concentration of metabolite BAY 1896953 characterized by Cmax | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  Cmax: maximum drug concentration in plasma after single dose administration
Plasma concentration of metabolite BAY 1896953 characterized by tmax | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  tmax: time to reach maximum drug concentration in plasma after single (first) dose
Plasma concentration of metabolite BAY 1896953 characterized by AUC(0-12) | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  AUC(0-12):AUC from time 0 to 12 hours after administration
Plasma concentration of diastereomers BAY 1896951 characterized by Cmax | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  Cmax: maximum drug concentration in plasma after single dose administration
Plasma concentration of diastereomers BAY 1896951 characterized by tmax | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  tmax: time to reach maximum drug concentration in plasma after single (first) dose
Plasma concentration of diastereomers BAY 1896951 characterized by AUC(0-12) | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  AUC(0-12):AUC from time 0 to 12 hours after administration
Plasma concentration of diastereomers BAY 1896952 characterized by Cmax | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  Cmax: maximum drug concentration in plasma after single dose administration
Plasma concentration of diastereomers BAY 1896952 characterized by tmax | tmax: time to reach maximum drug concentration in plasma after single (first) dose
  Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
Plasma concentration of diastereomers BAY 1896952 characterized by AUC(0-12) | Day -5 {pre dose, 0.5,1,1.5,3,5 ,8,12,24,36,48},Day -2 {before morning dose, 0.5,1,1.5,3,5,8, 12, 24, 36 and 48 h} ,Day 7 {before morning dose, 0.5, 1, 1.5,3,5,8,12 h (before evening dose)}
  AUC(0-12):AUC from time 0 to 12 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kashiwa, Chiba, Japan